CLINICAL TRIAL: NCT02907463
Title: Assessing Clinical Outcomes Using the EDWARDS INTUITY Elite Valve System in Isolated AVR Using Minimally InvaSive Surgery In a EurOpean Multi-ceNter, Active, Post-market Registry
Brief Title: EDWARDS INTUITY Elite Valve System
Acronym: MISSION
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015-05
Record Dates: First submitted 2016-06-29; First posted 2016-09-20 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Aortic Valve Disease; Aortic Stenosis
Keywords: Aortic Valve Replacement; Aortic Stenosis; EDWARDS INTUITY Elite; Rapid deployment valves
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this active, observational, open-label, non-randomized, post-market surveillance study is to confirm that EDWARDS INTUITY Elite reduces cross clamp time (XCT) in MIS setting when compared to published data with a conventional valve within the MIS setting. The published dataset will used as a control group. Then to describe short term (30 days) and long term (6 months) clinical safety, to assess and compare hemodynamic data with EDWARDS INTUITY Elite to a conventional valve at discharge and at 6 months post AVR, to assess Quality of Life at baseline, and at 6 months post AVR to assess NYHA functional class at baseline, discharge, 1 month and at 6 months post AVR to assess Fitness for hospital discharge.

DETAILED DESCRIPTION:
Aortic valve replacement with mechanical or biological heart valves is the treatment of choice for aortic valve stenosis. Over the past several years, life expectancy has increased in industrial nations, but this has been accompanied by a rising rate of elderly patients with multiple illnesses.

Aortic stenosis remains the most common cause of adult valvular heart disease, the prevalence increasing with age. Average survival of patients treated conservatively has historically been reported as 2-5 years from the onset of symptoms. More recent studies have confirmed the dismal prognosis of severe aortic stenosis. Advanced age, reduced left-ventricular ejection fraction, congestive heart failure and renal insufficiency appear to be independent predictors of reduced survival. Asymptomatic patients with very severe aortic stenosis also share a poor prognosis with a high event rate and a risk of rapid functional deterioration. Early surgery offers a therapeutic option to improve clinical outcomes via decreasing cardiac mortality and improving symptoms.

Bioprostheses offer several advantages over mechanical bioprostheses, the most important being freedom from anticoagulation with a low rate of thromboembolic accidents.

In response to clinical need and in support of advances in minimally invasive surgical approaches to conventional AVR, Edwards Lifesciences developed the EDWARDS INTUITY Elite Valve System to achieve clinical benefits by reducing cardiopulmonary bypass and cross clamp times, while facilitating a less invasive approach to aortic valve replacement.

The system includes the EDWARDS INTUITY Elite Valve System, Model 8300AB and the EDWARDS INTUITY Elite Delivery System, Model 8300DB; the valve is based on prior heart valve designs which have a long history of safety and effectiveness and have incorporated additional features designed to improve patient outcomes and safety.

With only 3 guiding sutures and secure balloon expandable frame, the EDWARDS INTUITY Elite Valve system is well suited for smaller incisions and tight access, with an emphasis on procedural efficiency within existing operating suite of the surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject is symptomatic for aortic stenosis (AS) or mixed aortic stenosis and aortic insufficiency (AS/AI) disease for which isolated surgical aortic valve replacement without concomitant procedures is indicated according to International guidelines.
3. Surgery starts with and is intended to be completed via a minimal invasive surgical approach. MIS is defined as a non-full sternotomy approach such as partial hemi-sternotomy, right anterior thoracotomy.
4. Surgery is intended to be completed with an EDWARDS INTUITY Elite Heart Valve.
5. Subject has signed and dated the investigation informed consent forms prior to any study-specific procedures are performed.
6. Subject is geographically stable and agrees to attend follow-up assessments as specified in the protocol and informed consent.

Exclusion Criteria:

1. Subject is diagnosed with pure aortic insufficiency.
2. Subject requires multiple valve replacement/repair
3. Subject has Type 0 congenital true bicuspid aortic valve (i.e. absence of raphe and commissures are positioned about 180 degrees apart) or unicuspid aortic valve.
4. Subject has severe ventricular dysfunction defined as LVEF < 25%.
5. Subject has a history of active endocarditis and/or myocarditis ≤ 3 months before the intended treatment/scheduled surgery.
6. Subject has had an acute MI ≤ 3 months before the intended treatment.
7. Subject had a stroke or transient ischemic attack within six months prior to scheduled aortic valve replacement surgery.
8. Subject is oxygen or ventilator dependent.
9. Subject has life expectancy < 12 months.
10. Female subject is pregnant or lactating.
11. Subject with documented leukopenia (WBC < 3.5x 103/μL), anemia (Hb < 10.0 gm/dL or < 6.2 mmol/L), thrombocytopenia (platelet count < 100x 103/mL), or history of bleeding diathesis or coagulopathy.
12. Subject has renal insufficiency as determined by Serum creatinine

    ≥ 200 μmol/L (2.27 mg/dL) at screening or end-stage renal disease requiring chronic dialysis.
13. Subject is currently participating in an investigational drug or device trial for which follow-up has not yet been completed.
14. Minimally Invasive access to the heart is not possible due to anatomical constraints or any other pre-existing condition.
15. Aneurysm of the aortic root and/or ascending aorta

Intra-operative exclusion criteria:

1. Subject has Type 0 congenital true bicuspid aortic valve (i.e. absence of raphe and commissures are positioned about 180 degrees apart) or unicuspid aortic valve. (A non-congenital bicuspid valve without a distorted annulus would not be cause for exclusion.)
2. Subject has calcium on the anterior mitral leaflet which cannot be removed.
3. Subject has extensive calcification of the aortic root.
4. Annular deformation which may or may not be caused by too extensive decalcification of the aortic annulus.
5. The position of the coronary ostia relative to the EDWARDS INTUITY Elite Aortic Valve could result in obstruction of blood flow.
6. Minimally Invasive access to the heart is not possible due to anatomical constraints or any other condition (including patient switched to a full sternotomy approach).
7. The device is not available in the correct size for the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult subjects, age18 or older, that have been diagnosed with aortic stenosis or stenosis-based insufficiency requiring isolated aortic valve replacement (AVR)
  * Subjects whose medical records indicate they are a suitable candidate for Minimally Invasive Surgery (MIS)
  * Subjects whose treating physician is the Principle Investigator or a Sub-Investigator participating in the study and has been trained on the EDWARDS INTUITY Elite Valve System
  * Subject shall be drawn from the general patient population served by each investigational center
  * Candidates for this study must meet all of the following Inclusion criteria and none of the Exclusion criteria or intra-op exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Young, MD FRCS, Principal Investigator — St. Thomas' Hospital; Gunther Laufer, Prof. Dr. med, Principal Investigator — AKH Vienna Dep. of Cardiovascular Surgery
Locations (23):
- Austria (2):
  - Universitätsklinik für Herzchirurgie Medizinische Universität Innsbruck, Innsbruck
  - Klinisshe Abteiluing Für Herz-thoraxchirurgie, Vienna
- Aarhus Universitets Hospital Skejby, Aarhus N, Denmark
- France (2):
  - CHU Bocage Central Dijon, Dijon
  - Hôpital Cardiologique CHU Bordeaux Haut Leveque, Pessac
- Germany (6):
  - Herz- und Gefäß-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale
  - Universitätsklinikum der Ruhr-Universität Bochum Klinik für Herz- und Thoraxchirurgie, Bochum
  - Herzzentrum Uniklinik Köln, Cologne
  - Medizinische Hochschule Hannover, Hanover
  - Herzzentrum Leipzig, Leipzig
  - University Hospital Würzburg, Würzburg
- Italy (5):
  - G. Pasquinucci Heart Hospital - "G.Monasterio" Foundation, Massa
  - CentroCardiologico Monzino, Milan
  - Clinica San Gaudenzio, Novara
  - Università Cattolica del Sacro Cuore Policlinico, Roma
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine
- Institut National de Chirurgie Cardiaque et Cardiologie Interventionnelle (INCCI), Luxembourg, Luxembourg
- St Antonius Hospital, Nieuwegein, Netherlands
- Spain (3):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Clínico San Carlos, Madrid
- United Kingdom (2):
  - Royal Infirmary Hospital Edinburgh, Edinburgh
  - St Thomas' Hospital, London

REFERENCES:
- [Derived] Laufer G, Strauch JT, Terp KA, Salinas M, Arribas JM, Massetti M, Andreas M, Young CP. Real-world 6-month outcomes of minimally invasive aortic valve replacement with the EDWARDS INTUITY Elite valve system. Interact Cardiovasc Thorac Surg. 2022 Jul 9;35(2):ivac083. doi: 10.1093/icvts/ivac083. PMID 35394527

RESULTS

PARTICIPANT FLOW:
Groups:
- EDWARDS INTUITY Elite Valve System: The system includes the EDWARDS INTUITY Elite Aortic Valve, Model 8300AB and the EDWARDS INTUITY Elite Delivery System, Model 8300DB.
Period: Overall Study
Arm/Group | EDWARDS INTUITY Elite Valve System
Started | 280
Enrolled Cohort | 280
Per Protocol Cohort | 276
Completed | 243
Not Completed | 37
Not completed — Lost to Follow-up | 17
Not completed — Death | 10
Not completed — Withdrawal by Subject | 4
Not completed — MIS Approach was not used | 2
Not completed — Not Implanted with Study Device | 2
Not completed — Device Explanted | 1
Not completed — Missing Exit Form | 1

BASELINE CHARACTERISTICS:
Groups:
- Per Protocol Cohort: The per protocol cohort will consist of all enrolled patients that leave the operating room with the registry valve in place and had an AVR MIS surgery procedure.
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 134
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subject's Average Time Spent on Cardiopulmonary Cross Clamp
Description: Cardiopulmonary cross clamp time is the amount of time that the patient's aorta (blood vessel) is clamped by a surgical instrument used in cardiac surgery. This allows the normal blood flow to be sent to an artificial heart and lung machine to keep it at a constant temperature and oxygen level.
Time Frame: At time of surgery; an average of 1 hour
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Per Protocol Cohort: The per protocol cohort consists of all enrolled patients that left the operating room with the registry valve in place and had an AVR MIS surgery procedure.
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
minutes
  Partial Sternotomy: number analyzed (Participants) | 240
  Partial Sternotomy | 49.9 (14.7)
  Right Thoracotomy: number analyzed (Participants) | 36
  Right Thoracotomy | 65.2 (18.2)
  All | 51.9 (16.0)

2. Secondary Outcome: Subject's Average Time Spent on Cardiopulmonary Bypass.
Description: Cardiopulmonary bypass time is the amount of time that the patient's blood circulates through an artificial heart and lung machine during cardiac surgery.
Time Frame: At time of surgery; an average of 1.5 hours
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
minutes | 79.0 (23.4)

3. Secondary Outcome: Device Technical Success Rate
Description: The successful delivery and deployment of the EDWARDS INTUITY Elite valve and delivery system, and the subject leaving the operating room with valve in place.
Time Frame: At time of surgery
Population: The outcome is reported for subjects where data is available. Analysis is based on the enrolled cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Cohort: A subject was considered enrolled into the registry when he/she signed the informed consent, and met all the registry eligibility criteria.
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 280
Participants | 276

4. Secondary Outcome: First Attempt Success Rate
Description: The successful delivery and deployment of the valve and delivery system during the first attempt, and subject leaving the operating room with EDWARDS INTUITY Elite valve in place.
Time Frame: At time of surgery
Population: The outcome is reported for subjects where data is available. Analysis is based on the enrolled cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 280
Participants | 270

5. Secondary Outcome: Procedural Success
Description: Procedural success is defined as device technical success followed by the absence of adverse events requiring device reoperation, requiring implantation of permanent pacemaker (with baseline sinus rhythm and no other conduction issues), or subject death, within discharge or 10 days post index procedure whichever comes first.
Time Frame: Day of procedure and events occurring within 10 days of procedure
Population: The outcome is reported for subjects where data is available. Analysis is based on the enrolled cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 280
Participants | 274

6. Secondary Outcome: Subject's Average Health Care Utilization
Description: The average amount of time the subjects spent in the intensive care unit and the average total length of hospital stay after their heart valve replacement procedure.
Time Frame: Day of surgical procedure through discharge from the hospital, an average of 3 days and 10 days respectively.
Population: The outcome is reported for subjects where data is available. Analysis is based on the enrolled cohort.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 278
days
  ICU Length of Stay: number analyzed (Participants) | 277
  ICU Length of Stay | 3.3 (7.2)
  Hospital Length of Stay | 9.5 (6.7)

7. Secondary Outcome: Subject's Average Mean Gradient Measurements Over Time.
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: Baseline, Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Per Protocol Cohort - 19mm; Per Protocol Cohort - 21mm; Per Protocol Cohort - 23mm; Per Protocol Cohort - 25mm; Per Protocol Cohort - 27mm; Per Protocol Cohort - Total: The per protocol cohort consists of all enrolled patients that left the operating room with the registry valve in place and had an AVR MIS surgery procedure.
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
mmHg
  Baseline: number analyzed (Participants) | 19 | 68 | 49 | 44 | 15 | 195
  Baseline | 50 (18.1) | 46.6 (13.7) | 44.5 (13.0) | 45.3 (13.4) | 45.1 (16.5) | 46.0 (14.1)
  Discharge: number analyzed (Participants) | 22 | 70 | 54 | 49 | 16 | 211
  Discharge | 15.0 (5.6) | 12.8 (5.0) | 9.7 (3.4) | 9.8 (3.6) | 7.6 (3.0) | 11.1 (4.7)
  6 months: number analyzed (Participants) | 23 | 65 | 51 | 44 | 16 | 199
  6 months | 11.7 (4.4) | 9.7 (3.4) | 8.0 (3.7) | 7.8 (2.6) | 6.1 (2.9) | 8.8 (3.7)

8. Secondary Outcome: Subject's Average Peak Gradients Measurements Over Time.
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: Baseline, Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
mmHg
  Baseline: number analyzed (Participants) | 19 | 68 | 49 | 44 | 15 | 195
  Baseline | 80.3 (25.9) | 78.9 (22.8) | 73.4 (20.8) | 74.8 (20.9) | 74.0 (22.0) | 76.3 (22.1)
  Discharge: number analyzed (Participants) | 22 | 70 | 54 | 49 | 16 | 211
  Discharge | 28.0 (10.4) | 25.0 (10.7) | 18.4 (6.6) | 18.6 (7.3) | 15.3 (6.2) | 21.4 (9.5)
  6 months: number analyzed (Participants) | 23 | 65 | 51 | 44 | 16 | 199
  6 months | 23.6 (8.4) | 19.7 (7.6) | 15.7 (6.7) | 15.0 (4.7) | 12.6 (4.9) | 17.5 (7.4)

9. Secondary Outcome: Subject's Average Effective Orifice Area (EOA) Measurements Over Time
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Baseline, Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
centimeters squared
  Baseline: number analyzed (Participants) | 17 | 61 | 47 | 40 | 12 | 177
  Baseline | 0.7 (0.2) | 0.8 (0.3) | 0.8 (0.2) | 0.9 (0.2) | 1.0 (0.2) | 0.8 (0.3)
  Discharge: number analyzed (Participants) | 21 | 54 | 42 | 41 | 14 | 172
  Discharge | 1.2 (0.3) | 1.5 (0.6) | 1.9 (0.6) | 2.0 (0.6) | 2.3 (0.7) | 1.8 (0.6)
  6 months: number analyzed (Participants) | 22 | 58 | 48 | 40 | 16 | 184
  6 months | 1.2 (0.3) | 1.5 (0.4) | 1.9 (0.5) | 2.1 (0.5) | 2.5 (0.6) | 1.8 (0.6)

10. Secondary Outcome: Subject's Average Effective Orifice Area Index (EOAI) Measurement Over Time.
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
centimeters squared/meters squared
  Discharge: number analyzed (Participants) | 18 | 44 | 36 | 38 | 14 | 150
  Discharge | 0.7 (0.2) | 0.9 (0.4) | 1.0 (0.3) | 1.0 (0.3) | 1.1 (0.4) | 0.9 (0.3)
  6 months: number analyzed (Participants) | 17 | 45 | 34 | 30 | 13 | 139
  6 months | 0.7 (0.1) | 0.8 (0.2) | 1.0 (0.3) | 1.1 (0.3) | 1.2 (0.3) | 0.9 (0.3)

11. Secondary Outcome: Subject's Average Performance Index Measurements Over Time.
Description: Performance index is defined as the subject's effective orifice area (the cross-sectional area of the blood flow downstream of the aortic valve) divided by the subject's pre-implant orifice area. Effective orifice area is evaluated by echocardiography over time.
Time Frame: Baseline, Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: cm2/cm2
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
cm2/cm2
  Baseline: number analyzed (Participants) | 17 | 61 | 47 | 40 | 12 | 177
  Baseline | 0.5 (0.1) | 0.5 (0.2) | 0.4 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 0.5 (0.2)
  Discharge: number analyzed (Participants) | 21 | 54 | 42 | 41 | 14 | 172
  Discharge | 0.9 (0.2) | 1.0 (0.4) | 1.0 (0.3) | 1.0 (0.3) | 0.9 (0.3) | 1.0 (0.3)
  6 months: number analyzed (Participants) | 22 | 58 | 48 | 40 | 16 | 184
  6 months | 1.0 (0.2) | 1.0 (0.2) | 1.0 (0.3) | 1.0 (0.2) | 1.0 (0.2) | 1.0 (0.2)

12. Secondary Outcome: Subject's Average Cardiac Output Over Time
Description: The amount of blood the heart pumps through the circulatory system in a minute.
Time Frame: Baseline, Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
liters per minute
  Baseline: number analyzed (Participants) | 17 | 61 | 45 | 40 | 10 | 173
  Baseline | 4.8 (1.2) | 5.3 (1.5) | 5.4 (1.3) | 6.1 (1.8) | 6.2 (1.5) | 5.5 (1.5)
  Discharge: number analyzed (Participants) | 21 | 53 | 41 | 41 | 13 | 169
  Discharge | 4.0 (1.1) | 4.9 (1.7) | 5.4 (1.5) | 5.7 (1.6) | 5.0 (1.4) | 5.1 (1.6)
  6 months: number analyzed (Participants) | 22 | 59 | 48 | 40 | 15 | 184
  6 months | 4.1 (0.9) | 4.5 (1.0) | 4.8 (1.4) | 5.2 (1.0) | 5.4 (1.6) | 4.8 (1.2)

13. Secondary Outcome: Subject's Average Cardiac Index
Description: A measure of cardiac output per square meter of body surface area
Time Frame: Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: L/min/meters squared
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
L/min/meters squared
  Discharge: number analyzed (Participants) | 18 | 43 | 36 | 38 | 13 | 148
  Discharge | 2.3 (0.6) | 2.7 (0.8) | 2.8 (0.8) | 2.8 (0.8) | 2.4 (0.7) | 2.7 (0.8)
  6 months: number analyzed (Participants) | 17 | 45 | 34 | 30 | 12 | 138
  6 months | 2.4 (0.3) | 2.5 (0.6) | 2.6 (0.9) | 2.6 (0.5) | 2.6 (0.6) | 2.6 (0.7)

14. Secondary Outcome: Subject's Amount of Paravalvular Leak Over Time.
Description: Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing. Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Count of Participants; unit: Participants
Groups:
- Per Protocol Cohort - All Subjects: The per protocol cohort consists of all enrolled patients that left the operating room with the registry valve in place and had an AVR MIS surgery procedure.
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - All Subjects
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
Participants
  Discharge: number analyzed (Participants) | 20 | 68 | 50 | 51 | 15 | 204
  Discharge: 0 None | 19 | 59 | 45 | 45 | 14 | 182
  Discharge: +1 Trivial/Trace | 1 | 6 | 5 | 5 | 0 | 17
  Discharge: +2 Mild | 0 | 3 | 0 | 1 | 0 | 4
  Discharge: +3 Moderate | 0 | 0 | 0 | 0 | 1 | 1
  Discharge: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  6 months: number analyzed (Participants) | 20 | 62 | 53 | 45 | 16 | 196
  6 months: 0 None | 18 | 55 | 49 | 40 | 15 | 177
  6 months: +1 Trivial/Trace | 1 | 6 | 4 | 4 | 0 | 15
  6 months: +2 Mild | 1 | 1 | 0 | 1 | 0 | 3
  6 months: +3 Moderate | 0 | 0 | 0 | 0 | 1 | 1
  6 months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Subject's Amount of Aortic Valvular Regurgitation Over Time.
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from minimum of 0 to maximum of 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge and 6 Months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Per Protocol Cohort - 19mm | Per Protocol Cohort - 21mm | Per Protocol Cohort - 23mm | Per Protocol Cohort - 25mm | Per Protocol Cohort - 27mm | Per Protocol Cohort - Total
Number analyzed (Participants) | 29 | 89 | 75 | 63 | 20 | 276
Participants
  Discharge: number analyzed (Participants) | 20 | 68 | 51 | 51 | 15 | 205
  Discharge: 0 None | 15 | 61 | 48 | 40 | 14 | 178
  Discharge: +1 Trivial/Trace | 5 | 7 | 3 | 11 | 1 | 27
  Discharge: +2 Mild | 0 | 0 | 0 | 0 | 0 | 0
  Discharge: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Discharge: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0
  6 months: number analyzed (Participants) | 20 | 62 | 54 | 45 | 16 | 197
  6 months: 0 None | 14 | 54 | 46 | 40 | 13 | 167
  6 months: +1 Trivial/Trace | 6 | 8 | 8 | 5 | 3 | 30
  6 months: +2 Mild | 0 | 0 | 0 | 0 | 0 | 0
  6 months: +3 Moderate | 0 | 0 | 0 | 0 | 0 | 0
  6 months: +4 Severe | 0 | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Subject's Average SF-36 Physical Health Summary
Description: The Medical Outcomes Study Short-Form 36 - Physical Health Summary The SF-36 questionnaire scale ranges from 100, which reflects the best health status to 0, which reflects the worse health status.
Time Frame: Baseline and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
units on a scale
  Baseline: number analyzed (Participants) | 209
  Baseline | 42.6 (8.1)
  6 months: number analyzed (Participants) | 209
  6 months | 47.6 (8.1)

17. Other Pre Specified Outcome: Subject's Average SF-36 Mental Health Summary
Description: The Medical Outcomes Study Short-Form 36 - Mental Health Summary The SF-36 questionnaire scale ranges from 100, which reflects the best health status to 0, which reflects the worse health status.
Time Frame: Baseline and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
units on a scale
  Baseline: number analyzed (Participants) | 209
  Baseline | 45.5 (10.4)
  6 months: number analyzed (Participants) | 209
  6 months | 50.1 (10.1)

18. Other Pre Specified Outcome: Subject's New York Heart Association (NYHA) Functional Class Compared to Baseline
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life. Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: 6 months compared to baseline
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 239
Participants
  Preoperative Classification, Class I: number analyzed (Participants) | 9
  Preoperative Classification, Class I: Class I | 9
  Preoperative Classification, Class I: Class II | 0
  Preoperative Classification, Class I: Class III | 0
  Preoperative Classification, Class I: Class IV | 0
  Preoperative Classification, Class II: number analyzed (Participants) | 111
  Preoperative Classification, Class II: Class I | 85
  Preoperative Classification, Class II: Class II | 25
  Preoperative Classification, Class II: Class III | 1
  Preoperative Classification, Class II: Class IV | 0
  Preoperative Classification, Class III: number analyzed (Participants) | 115
  Preoperative Classification, Class III: Class I | 71
  Preoperative Classification, Class III: Class II | 38
  Preoperative Classification, Class III: Class III | 6
  Preoperative Classification, Class III: Class IV | 0
  Preoperative Classification, Class IV: number analyzed (Participants) | 4
  Preoperative Classification, Class IV: Class I | 4
  Preoperative Classification, Class IV: Class II | 0
  Preoperative Classification, Class IV: Class III | 0
  Preoperative Classification, Class IV: Class IV | 0
  All Subjects: Class I | 169
  All Subjects: Class II | 63
  All Subjects: Class III | 7
  All Subjects: Class IV | 0

19. Other Pre Specified Outcome: Subject's Average Score on the EQ-5D - Quality of Life Questionnaire Over Time
Description: The EuroQol-5 Dimension (EQ-5D) is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline and 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
units on a scale
  Baseline: number analyzed (Participants) | 211
  Baseline | 0.73 (0.21)
  6 months: number analyzed (Participants) | 211
  6 months | 0.82 (0.22)

20. Other Pre Specified Outcome: Subject's Average Fitness for Hospital Discharge
Description: Considered as the day at which the patient was fit for hospital discharge.
Time Frame: Day of surgical procedure through discharge from the hospital; an average of 7 days
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 275
days | 6.8 (6.1)

21. Other Pre Specified Outcome: Number of Early Adverse Events Divided by Number of Subjects (Expressed as a Percentage)
Description: Number of early adverse events occurring within 30 days of procedure divided by the number of enrolled subjects times 100
Time Frame: Events occurring within 30 days of procedure
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Number; unit: Percentage of events/subjects
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
Percentage of events/subjects
  All Cause Mortality | 1.1
  Trial Valve Related Mortality | 0.0
  Thromboembolism | 3.6
  Stroke | 2.9
  TIA | 0.0
  Non-cerebral Embolism | 0.7
  Valve Thrombosis | 0.0
  Major Bleeding | 0.4
  Minor Paravalvular Leak (OPC) | 0.4
  Major Paravalvular Leak (OPC) | 0.4
  Hemolysis | 0.0
  NSVD Other than PVL | 0.0
  Endocarditis | 0.0
  Structural Valve Deterioration | 0.0
  Reoperation | 0.0
  Explant | 0.0
  Renal Failure | 2.2
  Respiratory Failure/Dysfunction | 1.1
  Deep Sternal Wound Infection | 0.7
  Permanent Pacemaker Implant | 6.7

22. Other Pre Specified Outcome: Number of Late Adverse Events Divided by Late Patient Years (Expressed as a Percentage)
Description: Number of late adverse events divided by the total number of late patient years x 100. Late patient years are calculated from 31 days post-implant to the date of the last contact (follow up or adverse event).
Time Frame: Events occuring >= 31 days and up through 6 months
Population: The outcome is reported for subjects where data is available. Analysis is based on the per protocol cohort.
Measure: Number; unit: percentage of events/late patient years
Arm/Group | Per Protocol Cohort
Number analyzed (Participants) | 276
percentage of events/late patient years
  All Cause Mortality | 6.1
  Trial Valve Related Mortality | 3.5
  Thromboembolism | 1.7
  Stroke | 1.7
  TIA | 0.0
  Non-cerebral Embolism | 0.0
  Valve Thrombosis | 0.0
  Major Bleeding | 2.6
  Minor Paravalvular Leak (OPC) | 0.0
  Major Paravalvular Leak (OPC) | 0.9
  Hemolysis | 0.0
  NSVD Other than PVL | 0.9
  Endocarditis | 0.0
  Structural Valve Deterioration | 0.9
  Reoperation | 1.7
  Explant | 1.7
  Renal Failure | 0.0
  Respiratory Failure/Dysfunction | 0.9
  Deep Sternal Wound Infection | 1.7
  Permanent Pacemaker Implant | 1.8

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through 6 months post implant
Description: This outcome is reported for subjects who received an EDWARDS INTUITY Elite Valve System where data is available.
Arm/Group | Per Protocol Cohort
All-Cause Mortality (participants affected / at risk) | 10/280
Serious Adverse Events (participants affected / at risk) | 108/280
Other Adverse Events (participants affected / at risk) | 155/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Cohort (N=280)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia - AV Block - 1st degree (Cardiac disorders) | 2 (2)
Arrhythmia - AV Block - 2nd degree (Cardiac disorders) | 2 (2)
Arrhythmia - AV Block - 3rd degree (Cardiac disorders) | 11 (11)
Arrhythmia - Atrial Flutter (Cardiac disorders) | 4 (4)
Arrhythmia - Bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - Bundle Branch Block - Left (Cardiac disorders) | 1 (1)
Arrhythmia - Other (Cardiac disorders) | 1 (1)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 16 (17)
Arrhythmia - Permanent Atrial Fibrillation (Cardiac disorders) | 1 (1)
Arrhythmia - Persistent Atrial Fibrillation (Cardiac disorders) | 7 (8)
Arrhythmia - Supraventricular Tachycardia (SVT) (Cardiac disorders) | 2 (2)
Arrhythmia - Tachy-Bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Biliary (Gallbladder) (Gastrointestinal disorders) | 1 (1)
Bleeding - Cardiovascular - Major (Blood and lymphatic system disorders) | 7 (7)
Bleeding - Gastrointestinal Lower - Minor (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Gastrointestinal Upper - Major (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Gastrointestinal Upper - Minor (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Neurological - Major (Blood and lymphatic system disorders) | 1 (1)
Bone Fracture / Break (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer - Newly diagnosed (General disorders) | 1 (1)
Cancer - Progression of underlying disease (General disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Chordae tendineae damage (Cardiac disorders) | 1 (1)
Deep Sternal Wound / Thoracic Infection (Infections and infestations) | 4 (4)
Fever - Unknown Origin (General disorders) | 2 (2)
Gastrointestinal - Infection (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 3 (3)
Hearing disorder (Ear and labyrinth disorders) | 1 (1)
Heart Failure - Acute (Cardiac disorders) | 7 (8)
Heart Failure - Chronic (CHF) (Cardiac disorders) | 1 (1)
Infection / Inflammation - Other (Infections and infestations) | 2 (2)
Multi-System organ failure (General disorders) | 1 (1)
Muscular Skeletal / Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
NSVD - LVOT damage (Cardiac disorders) | 1 (1)
NSVD - Paravalvular Leak - +2 (Cardiac disorders) | 2 (2)
Nonspecific, Unknown, or Other Body System - Other complication (General disorders) | 3 (3)
Pancreatic complication (Gastrointestinal disorders) | 1 (1)
Perforation - Atrial (Cardiac disorders) | 1 (1)
Pericardial Effusion - Major (Cardiac disorders) | 6 (6)
Pericardial Effusion - Minor (Cardiac disorders) | 1 (1)
Pericardial Tamponade (Cardiac disorders) | 10 (10)
Pleural Effusion - Bilateral (Cardiac disorders) | 4 (4)
Pleural Effusion - Left (Cardiac disorders) | 3 (4)
Pleural Effusion - Right (Cardiac disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Psychiatric - Other (Psychiatric disorders) | 1 (1)
Psychiatric Disorder (Psychiatric disorders) | 1 (1)
Pulmonary Embolism - Right (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Dysfunction (Renal and urinary disorders) | 1 (1)
Renal Failure - Acute (Renal and urinary disorders) | 4 (4)
Renal - Other (Renal and urinary disorders) | 1 (1)
Respiratory Failure - COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Failure - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Infection - Lower (Bronchitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Infection - Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Splenic complication (Blood and lymphatic system disorders) | 1 (1)
Sudden, Unexplained Death (General disorders) | 1 (1)
Superficial Wound Infection - Sternal (Infections and infestations) | 3 (3)
Thromboembolic Event - Other - Central - Hemiparesis (Cardiac disorders) | 2 (2)
Thromboembolic Event - Stroke (Cardiac disorders) | 8 (8)
Transient Psychotic Syndrome (Psychiatric disorders) | 3 (3)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1)
Vascular - Access Site Complication (Vascular disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Per Protocol Cohort (N=280)
Anemia - Bleeding related - Minor (Blood and lymphatic system disorders) | 7 (8)
Anemia - Non-bleeding related (Blood and lymphatic system disorders) | 13 (13)
Angina, Stable (Cardiac disorders) | 1 (1)
Arrhythmia - AV Block - 1st degree (Cardiac disorders) | 8 (8)
Arrhythmia - AV Block - 2nd degree (Cardiac disorders) | 1 (1)
Arrhythmia - AV Block - 3rd degree (Cardiac disorders) | 2 (2)
Arrhythmia - Atrial Flutter (Cardiac disorders) | 1 (1)
Arrhythmia - Bradycardia (Cardiac disorders) | 4 (4)
Arrhythmia - Bundle Branch Block - Left (Cardiac disorders) | 53 (53)
Arrhythmia - Bundle Branch Block - Right (Cardiac disorders) | 3 (3)
Arrhythmia - Paroxysmal Atrial Fibrillation (PAF) (Cardiac disorders) | 57 (59)
Arrhythmia - Paroxysmal Atrial Tachycardia (PAT) (Cardiac disorders) | 1 (1)
Arrhythmia - Persistent Atrial Fibrillation (Cardiac disorders) | 13 (13)
Arrhythmia - Tachy-Bradycardia (Cardiac disorders) | 1 (1)
Arrhythmia - Tachycardia - Non-Ventricular (Cardiac disorders) | 4 (5)
Arrhythmia - Tachycardia - Ventricular (Cardiac disorders) | 3 (3)
Arrhythmia - Ventricular Fibrillation (Cardiac disorders) | 1 (1)
Bleeding - Cardiovascular - Major (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Genitourinary - Major (Blood and lymphatic system disorders) | 1 (1)
Bleeding - Genitourinary - Minor (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Musculoskeletal/Dermatological - Minor (Blood and lymphatic system disorders) | 2 (2)
Bleeding - Pulmonary/Respiratory Minor (Blood and lymphatic system disorders) | 1 (1)
Blood/ Lymphatic - Other (Blood and lymphatic system disorders) | 2 (2)
Bone Fracture / Break (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiovascular - Other (Cardiac disorders) | 1 (1)
Endocrine complications (Endocrine disorders) | 1 (1)
Fever - Unknown Origin (General disorders) | 2 (2)
Gastrointestinal - Infection (Infections and infestations) | 1 (1)
Gastrointestinal - Other (Gastrointestinal disorders) | 2 (2)
Hepatic complication - Other (Hepatobiliary disorders) | 1 (1)
Hypertension - Pulmonary (Cardiac disorders) | 1 (1)
Hypertension - Systemic (Cardiac disorders) | 5 (5)
Hypotension (Cardiac disorders) | 1 (1)
Infection / Inflammation - Other (Infections and infestations) | 1 (1)
Metabolic complications (Metabolism and nutrition disorders) | 2 (2)
Muscular Skeletal / Dermatologic - Other (Musculoskeletal and connective tissue disorders) | 3 (3)
NSVD - Paravalvular Leak - +1 (Cardiac disorders) | 2 (2)
NSVD - Paravalvular Leak - +2 (Cardiac disorders) | 1 (1)
Nonspecific, Unknown, or Other Body System - Other complication (General disorders) | 5 (5)
Pericardial Effusion - Minor (Cardiac disorders) | 1 (1)
Pleural Effusion - Bilateral (Cardiac disorders) | 3 (3)
Pleural Effusion - Left (Cardiac disorders) | 4 (4)
Pleural Effusion - Right (Cardiac disorders) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Psychiatric - Other (Psychiatric disorders) | 4 (4)
Psychiatric Disorder (Psychiatric disorders) | 2 (2)
Pulmonary/Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Regurgitation - Aortic-Central/Transvalvular-+1 (Cardiac disorders) | 1 (1)
Renal Dysfunction (Renal and urinary disorders) | 7 (7)
Renal Failure - Acute (Renal and urinary disorders) | 6 (6)
Respiratory Infection - Lower (Bronchitis) (Infections and infestations) | 1 (1)
Respiratory Infection - Pneumonia (Infections and infestations) | 3 (3)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial Wound Infection - Sternal (Infections and infestations) | 3 (3)
Thrombocytopenia - Heparin Induced (HIT) (Blood and lymphatic system disorders) | 1 (1)
Transient Psychotic Syndrome (Psychiatric disorders) | 11 (11)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 6 (6)
Vascular - Access Site Complication (Vascular disorders) | 1 (1)
Vascular - Other (Vascular disorders) | 1 (1)
Wound Infection - Other (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation, but data analyses of site-specific results can occur only in intervals as specified in the CTA. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT02907463/Prot_SAP_ICF_000.pdf